CLINICAL TRIAL: NCT07028034
Title: Could the 6 Minute Step Test be Used Instead of the 6 Minute Walk Test to Assess Functional Capacity in Individuals With Chronic Low Back Pain?
Brief Title: The 6 Minute Step Test in Chronic Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2025-08/89
Record Dates: First submitted 2025-05-29; First posted 2025-06-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indıviduals with chronic low back pain

SUMMARY:
Our study aimed to investigate whether the 6 minute step test could be used as an alternative to the 6 minute walk test for assessing functional capacity in individuals with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic low back pain
* Chronic low back pain for at least the last 3 months
* Being aged 18-65
* Voluntary participation in the study

Exclusion Criteria:

* Having orthopedic or neurological impairments
* History of surgery due to chronic low back pain in the last 6 months
* Being pregnant
* Participating in regular physical activity in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic low back pain will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | 1st and 2nd day
  Functional capacity will be assessed with a 6 minute walk test and 6 minute step test, and total distance and total number of step will be recorded. Quadriceps muscle oxygenation will be assessed with a monitor during the tests.
Muscle function | 1st day
  will be evaluated with a 5 times sit to stand test and the total time recorded.

SECONDARY OUTCOMES:
Muscle strength | 1st day
  Hand grip and quadriceps femoris muscle strength will be evaluated with a dynamometer
Disability level | 1st day
  It will be assessed with Oswestry Disability Index. High scores (0-50 point) on the scale indicate the presence and severity of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)